CLINICAL TRIAL: NCT00003449
Title: Phase II Study of Weekly Paclitaxel and Gemcitabine in Platinum-Resistant Ovarian Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Platinum-Resistant Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066478 (5O-98-1); LAC-USC-5O981; NCI-G98-1460
Record Dates: First submitted 1999-11-01; First posted 2003-09-24 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Dexamethasone; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: dexamethasone
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of dexamethasone plus paclitaxel and gemcitabine in treating patients with platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, progression time, and survival of patients with platinum-resistant ovarian cancer treated with weekly paclitaxel and gemcitabine.
* Determine the toxic effects of this regimen in these patients.
* Evaluate the toxic effects and safety profile of premedication with steroids with this regimen in these patients.

OUTLINE: Patients are stratified according to prior treatment with paclitaxel (none or relapse more than 6 months after paclitaxel versus progressive disease or relapse less than 6 months after paclitaxel).

Patients receive dexamethasone IV, then paclitaxel IV followed by gemcitabine IV, for 3 consecutive weeks on days 1, 8, and 15. Treatment is continued every 4 weeks in the absence of disease progression or unacceptable toxicity.

All patients are followed until death.

PROJECTED ACCRUAL: Approximately 18-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent ovarian epithelial cancer
* Platinum resistant disease defined as:

  * Progression during the most recent platinum-based chemotherapy OR
  * Relapse less than 6 months after platinum-based chemotherapy
* Measurable or evaluable disease

  * Elevated CA-125 only allowed
  * Positive cytology only not eligible

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal (ULN)
* AST less than 3 times ULN

Renal:

* Creatinine no greater than 2 mg/dL

Neurologic:

* No peripheral neuropathy greater than grade 2

Other:

* No other serious medical illness or psychiatric conditions.

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent hematopoietic growth factors

Chemotherapy:

* See Disease Characteristics
* No prior gemcitabine
* No prior paclitaxel administered weekly

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Recovered from acute toxic effects secondary to prior therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 1998-05; Primary Completion 2002-06 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, MD, Study Chair — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States